CLINICAL TRIAL: NCT06990854
Title: Electroacupuncture for PHN: Efficacy and Biomarker Evaluation in a Multicenter, Randomized, Sham-Controlled Trial Protocol
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dexiong Han (Other Government)
Collaborators: The Third People's Hospital of Hangzhou (Other); Changxing County Traditional Chinese Medicine Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Dexiong Han, Chief Traditional Chinese Medicine Physician, Zhejiang Chinese Medical University
Organization: Zhejiang Chinese Medical University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZSLL-KY-2025-034
Record Dates: First submitted 2025-05-09; First posted 2025-05-25 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-04

CONDITIONS: Postherpetic Neuralgia ( PHN )
Keywords: acupuncture; Postherpetic Neuralgia; serum biomarkers; serum substance P; Neuropeptide Y
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Electroacupuncture; mecobalamin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Electroacupuncture group (Experimental): Acupoint prescription: The therapeutic protocol utilized Ashi points (localized to herpetic lesion areas) and Jiaji points (EX-B2, ipsilateral to affected dermatomes).
  Acupuncture procedure: For Ashi points, sterile disposable needles (0.25 mm diameter, 40 mm length) were inserted at a 15° angle to a depth of 15-20 mm, without deqi sensation or manual manipulation. For Jiaji points (EX-B2), needles (0.30 mm diameter, 50 mm length) were inserted perpendicularly to a depth of 40-45 mm, with twisting manipulation (90° rotation at 90 cycles/min) until patients felt soreness, numbness, or distension. Electroacupuncture was applied using the Hans-100A device, with dense-disperse wave mode (2/100 Hz) and intensity adjusted to patient tolerance, for 30 minutes.
  Pharmacological intervention: Identical to the pharmacotherapy group.
  Interventions: Device: Electroacupuncture (Hans-100A, Nanjing Jisheng Medical Technology, China); Drug: Pharmacotherapy：① Pregabalin ( Lyrica™ ，Pfizer Inc. America) ② Methylcobalamin ( Mecobalamin tablets， Weicai (China) Pharmaceutical Co., Ltd， China）
- Pharmacotherapy group (Active Comparator): In accordance with the Interpretation of the expert consensus on the whole-process management of herpes zoster-associated pain, patients received protocol-guided therapy consisting of: ① Pregabalin: Initial dose 75 mg twice daily. Dose may be titrated upward to 150 mg twice daily within one week based on therapeutic response and tolerability. Gradual discontinuation is recommended when clinically appropriate, tapered by 100 mg decrements every 3-7 days. ② Mecobalamin tablets: 5 mg three times daily.
  Interventions: Drug: Pharmacotherapy：① Pregabalin ( Lyrica™ ，Pfizer Inc. America) ② Methylcobalamin ( Mecobalamin tablets， Weicai (China) Pharmaceutical Co., Ltd， China）
- Sham acupuncture group (Sham Comparator): Acupoint prescription: Identical to the electroacupuncture group. Acupuncture procedure: The Streitberger needle, a widely reported placebo needle device in acupuncture RCTs, was applied for sham intervention. Blinding assessments have predominantly demonstrated successful masking outcomes. This telescoping blunt-tip needle achieves non-penetrating placebo stimulation through its retractable design. Its key advantage lies in evoking a skin-penetrating sensation akin to true needling through tissue compression, while avoiding actual dermal perforation to minimize specific therapeutic effects. Following the perception of needle insertion reported by patients, the device is retracted by approximately 1 mm and connected to electroacupuncture apparatus without electrical stimulation activation.
  Pharmacological intervention: Identical to the pharmacotherapy group.
  Interventions: Drug: Pharmacotherapy：① Pregabalin ( Lyrica™ ，Pfizer Inc. America) ② Methylcobalamin ( Mecobalamin tablets， Weicai (China) Pharmaceutical Co., Ltd， China）; Procedure: Streitberger Placebo Needle Set ( Asiamed )

INTERVENTIONS:
Device: Electroacupuncture (Hans-100A, Nanjing Jisheng Medical Technology, China) — Acupoint prescription: The therapeutic protocol utilized Ashi points (localized to herpetic lesion areas) and Jiaji points (EX-B2, ipsilateral to affected dermatomes).
  Acupuncture procedure: For Ashi points, sterile disposable needles (0.25 mm diameter, 40 mm length) were inserted at a 15° angle to a depth of 15-20 mm, without deqi sensation or manual manipulation. For Jiaji points (EX-B2), needles (0.30 mm diameter, 50 mm length) were inserted perpendicularly to a depth of 40-45 mm, with twisting manipulation (90° rotation at 90 cycles/min) until patients felt soreness, numbness, or distension. Electroacupuncture was applied using the Hans-100A device, with dense-disperse wave mode (2/100 Hz) and intensity adjusted to patient tolerance, for 30 minutes.
  Arms: Electroacupuncture group
Drug: Pharmacotherapy：① Pregabalin ( Lyrica™ ，Pfizer Inc. America) ② Methylcobalamin ( Mecobalamin tablets， Weicai (China) Pharmaceutical Co., Ltd， China） — Patients received protocol-guided therapy consisting of: ① Pregabalin: Initial dose 75 mg twice daily. Dose may be titrated upward to 150 mg twice daily within one week based on therapeutic response and tolerability. Gradual discontinuation is recommended when clinically appropriate, tapered by 100 mg decrements every 3-7 days. ② Methylcobalamin: 5 mg three times daily.
Procedure: Streitberger Placebo Needle Set ( Asiamed ) — The Streitberger needle, a widely reported placebo needle device in acupuncture RCTs, was applied for sham intervention. This telescoping blunt-tip needle achieves non-penetrating placebo stimulation through its retractable design. Its key advantage lies in evoking a skin-penetrating sensation akin to true needling through tissue compression, while avoiding actual dermal perforation to minimize specific therapeutic effects. Following the perception of needle insertion reported by patients, the device is retracted by approximately 1 mm and connected to electroacupuncture apparatus without electrical stimulation activation.
  Arms: Sham acupuncture group

SUMMARY:
The investigators are conducting a clinical study with the following objectives: to evaluate the clinical efficacy of electroacupuncture combined with pregabalin in treating Postherpetic Neuralgia(PHN); to investigate the correlation between serum biomarker levels and pain symptoms;and to determine whether serum biomarkers can serve as prognostic indicators for PHN.

This study utilizes a randomized controlled trial design with assessor blinding. A total of 207 eligible PHN patients were randomly assigned to three groups in a 1:1:1 ratio: the electroacupuncture group, the pharmacotherapy group, and the sham acupuncture group. Comparative analyses of pain intensity and serum biomarker concentrations were conducted across these groups.

For the assessment of clinical outcomes, the investigators employed the following measures: the Numerical Rating Scale(NRS), the Hamilton Anxiety Scale(HAMA), the Hamilton Depression Scale(HAMD), the 36-Item Short Form Health Survey(SF-36), serum levels of substance P(SP)and Neuropeptide Y(NPY), and inflammatory markers(IL-10,TNF-α). These assessments were performed at baseline and at the end of weeks 1, 2, 3, and 4 of treatment.

The investigators anticipate that this clinical trial will enhance our understanding of the therapeutic efficacy and underlying mechanisms of acupuncture in managing PHN. It aims to elucidate the relationship between serum biomarkers and the clinical manifestations of PHN, as well as to explore their potential prognostic value in disease outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for PHN;
* Age between 20 and 80 years old;
* Voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

* Pregnant or lactating women;
* Presence of severe liver or kidney dysfunction, malignant tumors, or other serious diseases;
* Presence of hematologic diseases or coagulation disorders;
* Presence of mental illness or other cognitive impairments, unable to understand or unwilling to cooperate with the study requirements.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Assessing the participants' pain intensity by the Numerical Rating Scale | Assessments were performed at baseline and at the end of weeks 1, 2, 3, and 4 of treatment.
  Pain intensity was assessed using the Numerical Rating Scale (NRS), an 11-point scale ranging from 0 ("no pain") to 10 ("intolerable pain"). This validated tool demonstrates rapid clinical utility and robust psychometric properties, including good reliability and validity in pain assessment.

SECONDARY OUTCOMES:
The number of pain episodes in the past 24 hours | Assessments were performed at baseline and at the end of weeks 1, 2, 3, and 4 of treatment.
  Daily documentation of pain episodes over 24-hour intervals to characterize symptom fluctuation patterns.
Psychological Status Assessment: Hamilton Anxiety Scale 36 ( HAMA ) | Assessments were performed at baseline and at the end of weeks 1, 2, 3, and 4 of treatment.
  Hamilton Anxiety Scale36 (HAMA): A 14-item clinician-administered tool evaluating anxiety severity across domains such as anxious mood, tension, and insomnia. Scores ≥14 indicate clinically significant anxiety.
Psychological Status Assessment: Hamilton Depression Scale37 (HAMD-21) | Assessments were performed at baseline and at the end of weeks 1, 2, 3, and 4 of treatment.
  Hamilton Depression Scale37 (HAMD-21): A 21-item instrument assessing core depressive symptoms spanning affective, cognitive, and somatic dimensions.
  Assessments were performed at baseline and at the end of weeks 1, 2, 3, and 4 of treatment.
The health-related quality of participants' life is assessed by The Short-Form 36 Health Survey | Assessments were performed at baseline and at the end of weeks 1, 2, 3, and 4 of treatment.
  The Short-Form 36 Health Survey (SF-36) quantified health-related quality of life across 8 domains (e.g., physical function, social role). This instrument has been extensively validated in chronic pain research.
Neuroregeneration Indicators: Neuropeptide Y (NPY) | Assessments were performed at baseline and at the end of weeks 1, 2, 3, and 4 of treatment.
  Neuropeptide Y (NPY) , a mediator of neuro-immune crosstalk and synaptic remodeling.
Neuroregeneration Indicators: Substance P (SP) | Assessments were performed at baseline and at the end of weeks 1, 2, 3, and 4 of treatment.
  Substance P (SP), a tachykinin modulating nociceptive signaling.
Inflammatory Markers : TNF-α | Assessments were performed at baseline and at the end of weeks 1, 2, 3, and 4 of treatment.
  TNF-α, a proinflammatory cytokine.
Inflammatory Markers : IL-10 | Assessments were performed at baseline and at the end of weeks 1, 2, 3, and 4 of treatment.
  IL-10, an anti-inflammatory cytokine.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yu Q, Wang X, Wu J, Zhang Q, Ying X, Ou L, Hu H, He K, Wu L, Jin Z, Shentu J, Dai H, Ma R, Hu Q, Han D. Efficacy and Safety of Electroacupuncture for Postherpetic Neuralgia and Biomarker Evaluation: A Study Protocol for a Multicenter, Randomized Trial. J Pain Res. 2025 Nov 1;18:5753-5768. doi: 10.2147/JPR.S559309. eCollection 2025. PMID 41199896